CLINICAL TRIAL: NCT02022514
Title: Phase III Clinical Trial, Multicentric, Open, Randomized and Controlled to Assess the Effectiveness of Intracoronary Infusion of Mononuclear Cells Autologous Bone Marrow in Patients With Chronic Coronary Occlusion and Ventricular Dysfunction, Previously Revascularized.
Brief Title: Intracoronary Infusion of Mononuclear Cells Autologous Bone Marrow in Patients With Chronic Coronary Occlusion and Ventricular Dysfunction, Previously Revascularized.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMMo/OCC/2012
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Coronary Atherosclerosis and Other Heart Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mononuclear cells from autologous bone marrow (Experimental): Mononuclear bone marrow cells autologous intracoronary
  Interventions: Other: Mononuclear cells from autologous bone marrow
- Conventional medical treatment (Active Comparator): Conventional medical treatment
  Interventions: Drug: Conventional medical treatment

INTERVENTIONS:
Other: Mononuclear cells from autologous bone marrow — Mononuclear bone marrow cells autologous intracoronary
  Arms: Mononuclear cells from autologous bone marrow
Drug: Conventional medical treatment
  Arms: Conventional medical treatment

SUMMARY:
Clinical trial phase III, prospective, controlled, randomized, open.

We hypothesize work that patients with chronic coronary occlusion and poor myocardial viability who failed to recover ventricular function after subjecting coronary revascularization with new techniques of recanalization, could achieve an improvement of ventricular function if given further regenerative treatment with mononuclear cells from autologous bone marrow.

To test this hypothesis we designed a prospective, randomized clinical trial in patients with recanalized chronic occlusions and ventricular dysfunction.

DETAILED DESCRIPTION:
This is a randomized, open label prospective clinical trial in which all patients diagnosed with chronic coronary occlusion in the Cardiology Department of Hospital Reina Sofía in Cordoba and Hospital Puerta del Mar in Cadiz, who meet inclusion criteria and none of the exclusion shall include and express their accordance with trial participation by signing the informed consent.

66 patients who did not improve ventricular function measured by Magnetic resonance at least 3 months after revascularization of chronic coronary occlusion will be included . The 66 patients will be randomized in one to one ratio to an intervention group that received bone marrow mononuclear cells by intracoronary autologous (0.5 to 1 x 10 9 total cells) and a control group who receive only conventional medical treatment. The two groups of patients will be followed, in the clinical trial, for 6 months. Once the test is complete, they will follow according to standard clinical practice of Cardiology hospital for at least 24 months.

Patients will be assessed by clinical and Magnetic resonance methods. All patients will be medically treated similarly with ACE inhibitors or angiotensine 1 receptor (AT1) receptor antagonists of angiotensin II, beta-blockers and diuretics.

The main objective os the study is to determine the efficacy of intracoronary infusion of mononuclear cells from autologous bone marrow in patients with chronic coronary occlusion previously revascularized with stents in terms of improved ventricular function determined by magnetic resonance.

Secondary objectives of the study are:

1. To confirm, in view of the obtained results, the suitability of the proved protocol for the treatment of chronic coronary occlusion.
2. To study changes in functional class (I-IV NYHA) of these patients compared with the control group.
3. To evaluate the safety of treatment, the analysis of possible cardiac events during the 6-month follow-up in the clinical trial and 24 months of additional clinical follow-up (death, myocardial infarction, repeat revascularization) compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who give their informed consent to participate in this clinical trial.
2. Patients of both sexes with atherosclerotic coronary artery disease and chronic occlusions that recanalization has been achieved successfully implanted medicated stents, and in which nevertheless persists ventricular dysfunction evaluated by magnetic resonance.
3. Aged between 18 and 80 years.
4. Magnetic resonance performed at least 3 months of recanalization, the ejection fraction patient should remain below or iqual to 45%.
5. Normal renal function or mild renal insufficiency with serum creatinine exceeding 2.5 mg / dl.
6. Normal hepatic transaminases values function < 2,5 times the upper limit of the normal range.
7. Hemogram and coagulation studies were within normal values, defined by:

   * Leucocytes ≥ 3000
   * Neutrophils ≥ 1500
   * Platelets ≥ 100000
   * Hemoglobin > 10g/dl
8. Blood pregnancy test with negative results in the case of patients of childbearing age.
9. Acceptance by patients (both men and women) of childbearing age to use safe contraceptive methods throughout the study, including the six month follow-up.
10. Willingness and ability to implement the program of visits, treatment plan, laboratory tests, and all study procedures.

Exclusion Criteria:

1. Patients with chronic occlusions that recanalization were not achieved successfully.
2. Patients with ejection fractions upper to 45% after 3 months of recanalization.
3. Positive serology for HIV, HCV or HBV.
4. Coexistence of other serious systemic diseases or contraindication for double antiaggregation (clopidogrel and aspirin).
5. Coexistence of any type of hematological disease.
6. Pregnant, breast-feeding, or women of childbearing age who are not using effective contraception. A woman of childbearing age is considered to be all women from the age of 18 and up to one year after the last menstruation in the case of menopausal women.
7. Patients who are currently participating or have completed their participation in a clinical trial within a period of less than 3 months or who have participated in a clinical trial of Advanced Therapies (cell therapy, gene therapy or tissue engineering) at any time before and has been assigned to an experimental group.
8. Patients with malignant or pre-malignant tumors.
9. Patients in whom an MRI cannot be performed because they carry devices incompatible with the MRI (prostheses, defibrillators, pacemakers, etc).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the change in ejection fraction measured by magnetic resonance between inclusion and at 6 months follow-up | 6 months

SECONDARY OUTCOMES:
Changes of NYHA functional grade comparative manner between the groups. | 6 months
Possible cardiac events during follow-up (death, myocardial infarction, repeat revascularization). | 6 months
Need for hospital admission or presence of major arrhythmia | 6 months
Changes in global and segmental left ventricular function | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauel Pan Álvarez-Ossorio, MD, PhD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (2):
- Spain (2):
  - Dr. Alejandro Gutierrez, Cadiz
  - Hospital U. Reina Sofía, Seville